CLINICAL TRIAL: NCT04137575
Title: A Randomized Controlled Trial of ConquerFear: A Group-Based Psychological Intervention for Fear of Cancer Recurrence in Cancer Survivors
Brief Title: ConquerFear-Group: A Psychological Intervention for Fear of Cancer Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Nina M. Tauber, MSc, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NINTAU
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Fear of Cancer Recurrence; Breast Cancer Female
Keywords: Fear of Cancer Recurrence; Cancer Survivorship; Breast Cancer; Distress; Emotion Regulation
MeSH Terms: conditions — Breast Neoplasms; Emotional Regulation | interventions — Relaxation Therapy

STUDY DESIGN:
Intervention Model Description: Participants are randomized in blocks of 16. Participants in each block will be randomly assigned in a 1:1 ratio to either CF-G or CC, resulting 2 x 8 groups of approx. 8 participants (min 5 and max 10 participants in each group). A computer-generated randomization list will be created by a person not directly involved in the intervention. Allocation to condition will take place after completion of the baseline questionnaire package
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator and assessor is masked in terms of not knowing to which condition the participants will be randomized until after completion of the baseline assessment. The participants are masked in terms of not knowing that one intervention is hypothesized to yield larger effects than the other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ConquerFear-Group (Experimental): ConquerFear-Group is a psychological intervention developed specifically for fear of cancer recurrence
  Interventions: Behavioral: ConquerFear-Group
- Relaxation Training (Placebo Comparator): The Relaxation Training serves as a placebo comparator and is not developed specifically to target fear of cancer recurrence.
  Interventions: Behavioral: Relaxation Training

INTERVENTIONS:
Behavioral: ConquerFear-Group — The intervention consist of one 1½-hour individual session in which a psychologist will conduct an oral psychological assessment, and five 2-hour group sessions. The key goals of the intervention are to: a) teach strategies for controlling worry and excessive threat monitoring; b) modify underlying unhelpful beliefs about worry; c) develop appropriate monitoring and screening behaviors; d) educate about follow-up care and empirically-supported behavioral change (e.g., weight loss, exercise, etc.) to improve overall survival; e) address existential changes brought about by a cancer diagnosis; f) promote goal-setting. Each session is accompanied by home-based practice of skills learned in session and home reading to consolidate skill acquisition. Four trained psychologists (MSc) will perform the therapy. The intervention will be delivered on Zoom, a secure online platform.
  Arms: ConquerFear-Group
Behavioral: Relaxation Training — The control group will receive one 1½-hour individual session and participate in five 2-hour group sessions. Patients will receive guided progressive muscle relaxation training. The intervention will be delivered on Zoom, a secure online platform.
  Arms: Relaxation Training

SUMMARY:
The primary aim of this randomized controlled trial is to evaluate the effect of ConquerFear-Group (CF-G), compared with a control condition (CC), on Fear of Cancer Recurrence (FCR). Secondary aims are to explore the effect of CF-G on emotion regulation and additional psychological outcomes, and to explore mediating effects of emotion regulation, metacognitions, working alliance, patient adherence, and group cohesion. In addition, treatment expectancy, participation in other treatments after completion of the intervention of the study and demographic and clinical variables will be explored as moderators.

DETAILED DESCRIPTION:
A randomized controlled trial testing the efficacy of ConquerFear-Group (CF-G) on breast cancer survivors with clinical levels of Fear of Cancer Recurrence (FCR), compared with a control condition (CC), will be conducted.

The aims are to:

1. Evaluate the efficacy of CF-G on FCR,
2. Explore the effects on the secondary outcomes of emotion regulation, general distress, health-related QoL, survivors' unmet needs, mindfulness, metacognitions, intervention satisfaction, negative effects of intervention, and sleep.
3. Explore emotion regulation, metacognitions, working alliance, patient adherence, and group cohesion will be explored as possible mediators.*
4. Explore treatment expectancy, participation in other treatments after completion of the CF-G or the CC and demographic and clinical variables as possible moderators.

Primary hypothesis:

CF-G will yield larger reductions in FCR than CC at post treatment, and the effect will be maintained through the follow-up period.

Secondary hypotheses:

CF-G will demonstrate a larger improvement in measures of emotion regulation than CC following the intervention period.

Changes in emotion regulation during treatment will mediate the effect of CF-G on FCR.* Changes in metacognitions during treatment will mediate the effect of CF-G on FCR.* CF-G will yield larger reductions in general distress, health-related QoL, survivors' unmet needs than CC, and CF-G will yield larger improvements in metacognitions, mindfulness, and sleep than CC following the intervention period.

*The prerequesties for conducting for mediation analysis were not fulfilled. Consequently, these analyses were abandoned. Data can be obtained upon request.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients have a confirmed past diagnosis of stage 1-3 breast cancer,
2. have been treated with curative intent,
3. have completed all hospital-based adjuvant treatments 3 months to 5 years prior to study entry,
4. are disease free,
5. scores in the clinical range (≥22) on the Short Form of the Fear of Cancer Recurrence Inventory (FCRI-SF),
6. are able to read and write Danish,
7. are over the age of 18 years, and
8. are able to give informed consent.

Exclusion Criteria:

1. self-reported current major depression,
2. currently receiving psychological treatment from a therapist not involved in the study,
3. self-reported active psychotic illness or other severe psychiatric conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Fear of cancer recurrence | Baseline, 1, 2, 3, 4, 5, and 6 weeks after baseline, 1 week post intervention, 3- and 6-months follow-up
  Changes in fear of cancer recurrence will be measured with the 42-item Fear of Cancer Recurrence Inventory at baseline, 1 week post intervention, 3- and 6-months follow-up, and session-by-session with the 9-item Fear of Cancer Recurrence Inventory-Short Form

SECONDARY OUTCOMES:
Emotion regulation | Baseline, one week post intervention, 3- and 6-months follow-up
  Changes in emotion regulation will be assessed with the Difficulties in Emotion Regulation Questionnaire
General distress 1 | Baseline, one week post intervention, 3- and 6-months follow-up
  Changes in general distress will be measured with the Impact of Event Scale-Revised Questionnaire
General distress | Baseline, one week post intervention, 3- and 6-months follow-up
  Changes in general distress will be measured with the Depression, Anxiety, Stress Scale-21 Questionnaire
Health-related quality-of-life | Baseline, one week post intervention, 3- and 6-months follow-up
  Changes in health-related quality-of-life will be measured with the European Organization for Research and Treatment of Cancer QLQ-C30 Questionnaire
Health-related quality-of-life | Baseline, one week post intervention, 3- and 6-months follow-up
  Changes in health-related quality-of-life will be measured with EuroQol-5 Domain Questionnaire
Survivors' unmet needs | Baseline, one week post intervention, 3- and 6-months follow-up
  Changes in survivors' unmet needs will be measured with the Survivors' Unmet Need Survey - 8 item Information Sub-Scale Questionnaire
Fear of cancer recurrence | Baseline, one week post intervention, 3- and 6-months follow-up
  Changes in fear of cancer recurrence will be measured with the Concerns About Recurrence Questionnaire
Metacognitions | Baseline, one week post intervention, 3- and 6-months follow-up
  Changes in metacognitions will be measured with the Metacognitions Questionnaire-30
Mindfulness | Baseline, one week post intervention, 3- and 6-months follow-up
  Changes in mindfulness will be measured with the Five Facet Mindfulness Questionnaire
Sleep | Baseline, one week post intervention, 3- and 6-months follow-up
  Changes in sleep will be measured with the Insomnia Severity Index
Negative effects of intervention | One week post intervention, 3- and 6-months follow-up
  Negative effects of the intervention will be assessed with one question about negative effects of the intervention experienced by the participants (narrative response)
Negative effects of intervention | One week post intervention, 3- and 6-months follow-up
  Negative effects of the intervention will be measured with the Negative effects Questionnaire - hopelessness and failure subscales
Intervention satisfaction | One week post intervention, 3- and 6-months follow-up
  Intervention satisfaction will be measured with three questions regarding satisfaction with the treatment

OTHER OUTCOMES:
Moderator: Background information about the participants | Assessed at baseline only
  Background information about the participants will be assessed with a questionnaire regarding demongraphic information as possible moderators
Moderator: Clinical data | Collected from patients records
  Clinical data will be explored as possible moderators
Moderator: Treatment expectancy | Assessed at baseline only
  Treatment expectancy will be measured with the Credibility/Expectancy questionnaire as a possible moderator
Participation in other psychological, medical or complementary and alternative treatments for FCR after completion of the interventions of the present study | Assessed at 3- and 6-months follow-up
  Two questions regarding participation in other psychological, medical or complementary and alternative treatments for FCR after completion of the interventions of the present study will be assessed as a possible moderator
Mediator: Emotion regulation | Assessed 1, 2, 3, 4, 5, and 6 weeks after baseline.
  Changes in emotion regulation will be measured with the Brooding - Rumination and Reflection Scale
Mediator: Emotion regulation | Assessed 1, 2, 3, 4, 5, and 6 weeks after baseline.
  Changes in emotion regulation will be measured with the Penn State Worry Questionnaire
Mediator: Emotion regulation | Assessed 1, 2, 3, 4, 5, and 6 weeks after baseline.
  Changes in emotion regulation will be measured with the Experience Questionnaire
Mediator: Metacognitions | Assessed 1, 2, 3, 4, 5, and 6 weeks after baseline.
  Changes in metacognitions will be measured with the Metacognitions Questionnaire-30
Mediator: Working alliance | Assessed 1, 2, 3, 4, 5, and 6 weeks after baseline.
  Changes in working alliance will be measured with the Working Alliance Inventory Revised Short Form
Mediator: Patient adherence | Assessed 3, 4, 5, and 6 weeks after baseline.
  Changes in patient adherence will be assessed with a diary of home exercise completion
Mediator: Group cohesion | Assessed 2, 3, 4, 5, and 6 weeks after baseline.
  Changes in group cohesion will be assessed with the Therapeutic Factors Inventory Cohesiveness Scale
Mediator: Level of physical relaxation/calmness | Assessed 1, 2, 3, 4, 5, and 6 weeks after baseline.
  Single question to asses level of physical relaxation before and after each session
Mediator: Level of mental calmness | Assessed 1, 2, 3, 4, 5, and 6 weeks after baseline.
  Single question to asses level of mental calmness before and after each session

CONTACTS AND LOCATIONS:
Overall Officials: Robert Zachariae, DMSc, Study Director — Department of Oncology, Aarhus University Hospital & Aarhus University
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All data underlying publication will be shared in accordance with current data sharing regulations at host institutions.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: Researchers aiming to publish IPD meta-analyses. The authors to review requests are the PI and senior supervisors (NT, MSO, RZ, PB).